CLINICAL TRIAL: NCT06282497
Title: Xerostomia-optimised Intensity-modulated Radiotherapy Versus Standard Intensity-modulated Radiotherapy in Nasopharyngeal Carcinoma Patients:a Multicenter Non-inferior Randomized Controlled Phase III Clinical Trial
Brief Title: Xerostomia-optimised IMRT Versus Standard IMRT in NPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Gui-Qiong Xu, Chief Physician, Zhongshan People's Hospital, Guangdong, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSCPH-003
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-02

CONDITIONS: Nasopharyngeal Carcinoma ,Xerostomia,Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): optimised neck CTV delineation
  Interventions: Radiation: Optimised neck CTV
- Control Group (Active Comparator): standard neck CTV delineation
  Interventions: Radiation: standard neck CTV

INTERVENTIONS:
Radiation: Optimised neck CTV — neck CTV delineation extends from the lateral process of C1
  Arms: Study Group
Radiation: standard neck CTV — neck CTV delineation extends from skull base
  Arms: Control Group

SUMMARY:
This is a multi-center, non-inferiority, open-label, randomized controlled phase III clinical trial in primary diagnosed nasopharyngeal carcinoma (NPC) patients without distant metastasis. This study aims to compare the regional control, survival outcomes, radiation-related toxicities, and quality of life (QoL) of xerostomia-optimized intensity-modulated radiotherapy versus standard intensity-modulated radiotherapy in NPC patients

DETAILED DESCRIPTION:
Xerostomia remains one of the most common radiation-induced toxicities, and approximately 80% to 90% of NPC patients still experience varying degrees of xerostomia post-IMRT. Among the major salivary glands, the parotid gland is the largest and produces 60% to 65% of the oral saliva output. Studies have revealed that xerostomia post-IMRT is mainly dependent on the irradiation dose of the parotid glands. Clinical target volumes (CTV) for the cervical nodal region starting from skull base have been the standard in nasopharyngeal carcinoma for several decades. Consequently, the parotid glands overlap with the target volumes and irradiation dose reaches 31.7 Gy to 43.9 Gy in most reports. Retrospective studies reveal that the lateral process of C1 is a suitable cranial edge for neck CTV delineation; therefore, the volume of the parotid glands exposed to high radiation doses can be greatly reduced. we conducted this trial comparing outcomes ,toxicities and QoL of xerostomia-optimized intensity-modulated radiotherapy versus standard intensity-modulated radiotherapy in nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal non-keratinizing carcinoma (WHO II/III);
* All genders, range from 18-70 years old;
* ECOG score 0-1;
* Clinical stage I-IVa (AJCC/UICC 8th);
* Not received radiotherapy, chemotherapy and other anti-tumor treatment (including immunotherapy);
* No contraindications to chemotherapy or radiotherapy;
* Adequate organ function: white blood cell count ≥ 4×109/L, neutrophile granulocyte count ≥ 1.5×109/L, hemoglobin ≥ 90g/L, platelet count ≥ 100×109/L; alanine aminotransferase or aspartate aminotransferase < 2.5×upper limit of normal; blood urea nitrogen or creatinine ≤ 1.5×upper limit of normal or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Sign the consent form.

Exclusion Criteria:

* Level II involvement with extracapsular extension (ECE), and/or had a maximum nodal axial diameter (MAD) of greater than 3cm in level II ;

  -≥4 nodal regions of ipsilateral neck involvement;
* Radiologically suspicious or confirmed involvement in level II area between skull base and the lateral process of C1;
* Parotid lymph node and/or parotid gland involvement;
* History of parotid disease or surgery;
* Previous malignancy or other concomitant malignant disease;
* Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2029-10-23 (Estimated)

PRIMARY OUTCOMES:
Regional recurrence free survival | 3 years
  From the date of randomization to regional recurrence or any death

SECONDARY OUTCOMES:
Overall survival | 3 years
  From the date of randomization to any death, with patients unavailable for follow-up censored at the date of last follow-up
Local recurrence free survival | 3 years
  From the date of randomization to local recurrence or any death
Distant metastasis-free survival | 3 years
  From the date of randomization to distant metastasis or any death
Progression free survival | 3 years
  From the date of randomization to local or regional recurrence, distant metastasis or any death
Acute toxicities | From the start of treatment until 3 months post treatment
  Assessed with CTCAE v5.0
Late toxicities | 3 years post treatment
  Assessed with Radiation Therapy Oncology Group criteria and the CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gui-qiong Xu, MD, Principal Investigator — Zhongshan People's Hospital, Guangdong, China
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China